CLINICAL TRIAL: NCT00301964
Title: A Phase II Evaluation of Bevacizumab (NCI-Supplied Agent: NSC# 704865, IND # 7921) in the Treatment of Recurrent or Persistent Endometrial Carcinoma
Brief Title: Bevacizumab in Treating Patients With Recurrent or Persistent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02692; NCI-2012-02692 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000465502; GOG-0229E (Other: Gynecologic Oncology Group); GOG-0229E (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Recurrent Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Bevacizumab

ARMS (1):
- Treatment (bevacizumab) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well bevacizumab works in treating patients with recurrent or persistent endometrial cancer. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the activity of bevacizumab, in terms of 6-month progression-free survival rate and objective tumor response, in patients with recurrent or persistent endometrial cancer.

II. Determine the nature and degree of toxicity of bevacizumab in these patients.

SECONDARY OBJECTIVES:

I. Determine the duration of progression-free survival and overall survival of these patients.

II. Determine the effects of prognostic factors, including performance status and histological grade.

OUTLINE:

Patients receive bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or persistent endometrial carcinoma with histologic confirmation of the original primary tumor

  * Refractory to curative therapy or established treatments
* Measurable disease

  * At least one non previously irradiated lesion that can be accurately measured in ≥ 1 dimension as ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan

    * Previously irradiated lesion allowed provided disease progression is documented or a biopsy obtained to confirm persistent disease ≥ 90 days after completion of prior radiotherapy
* Must have received 1 prior chemotherapy regimen for endometrial carcinoma

  * May include high-dose therapy, consolidation, or extended therapy after surgical or nonsurgical assessment
* Not eligible for a higher priority GOG protocol, if one exists
* No tumor involving major vessels
* No prior history or evidence of CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy, or any brain metastases
* GOG performance status (PS) 0-2 (if received 1 prior treatment regimen)
* GOG PS 0-1 (if received 2 prior treatment regimens)
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Serum bilirubin ≤ 1.5 times ULN
* SGOT and alkaline phosphatase ≤ 2.5 times ULN
* Urine protein:creatinine ratio < 1.0
* INR < 1.5 (or in-range, usually between 2 and 3, if the patient is on a stable dose of therapeutic warfarin)
* PTT < 1.5 times ULN
* No active infection requiring antibiotics
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study therapy
* No serious nonhealing wound or ulcer, including any of the following:

  * History of abdominal fistula
  * Gastrointestinal perforation
  * Intra-abdominal abscess within the past 28 days
* No serious nonhealing bone fracture
* No active bleeding or pathologic conditions that carry high risk of bleeding, including known bleeding disorder or coagulopathy
* No clinically significant cardiovascular disease, including any of the following:

  * Uncontrolled hypertension, defined as systolic blood pressure (BP) > 150 mm Hg or diastolic BP > 90 mm Hg
  * Myocardial infarction or unstable angina within the past 6 months
  * New York Heart Association class II-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Ejection fraction < 50% and received prior anthracycline (including doxorubicin and/or doxorubicin HCl liposomal)
  * Grade 2 or greater peripheral vascular disease
  * History of cerebrovascular accident, transient ischemic attack, or subarachnoid hemorrhage within the past 6 months
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
* No significant traumatic injury within the past 28 days
* See Disease Characteristics
* Recovered from recent surgery, radiotherapy, or chemotherapy
* Hormonal therapy directed at the malignant tumor must be discontinued ≥ 1 week prior to registration
* Any other prior therapy directed at the malignant tumor, including immunologic agents, must be discontinued ≥ 3 weeks prior to registration
* No prior chemotherapy or radiotherapy to any portion of the abdominal cavity or pelvis

  * Prior chemotherapy or radiotherapy for localized cancer of the breast, head and neck, or skin for which the patient remains free of recurrent or metastatic disease is allowed provided it was completed ≥ 3 years prior to study
* No prior cancer treatment that contraindicates study therapy
* No prior bevacizumab or other vascular endothelial growth factor (VEGF) pathway-targeted therapy
* One additional prior cytotoxic regimen for recurrent or persistent endometrial cancer allowed, including any agent that targets the genetic and/or mitotic apparatus of dividing cells resulting in dose-limiting toxicity to the bone marrow and/or gastrointestinal mucosa
* No prior noncytotoxic chemotherapy for recurrent or persistent disease
* More than 28 days since major surgical procedure or open biopsy
* More than 7 days since minor surgical procedures, fine needle aspirates, or core biopsies
* No concurrent major surgical procedure
* No concurrent prophylactic filgrastim (G-CSF) or thrombopoietic agents
* No concurrent amifostine or other protective reagents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Aghajanian, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Bevacizumab)
Started | 56
Completed | 52 (Total number of eligible and evaluable participants)
Not Completed | 4
Not completed — Second primary | 2
Not completed — Wrong primary | 1
Not completed — Inadequate pathology | 1

BASELINE CHARACTERISTICS:
Population: Total number of eligible and evaluable participants
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (10.3)
Age, Customized [Number; unit: participants]
  30-39 years | 1
  40-49 years | 4
  50-59 years | 13
  60-69 years | 22
  70-79 years | 11
  80-89 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 52
Cell Type [Number; unit: participants]
  Adenocarcinoma, Unspecified | 1
  Clear Cell Carcinoma | 4
  Endometrioid Adenocarcinoma | 26
  Mucinous Adenocarcinoma | 1
  Mixed Epithelial Carcinoma | 5
  Undifferentiated Carcinoma | 1
  Serous Adenocarcinoma | 14

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Greater Than 6 Months
Description: Disease Progression is at least a 20% increase in the sum of longest dimension (LD) of target lesions taking as references the smallest sum LD or the appearance of new lesions within 8 weeks of study entry.
Time Frame: 6 months
Population: Total number of eligible and evaluable participants
Measure: Number; unit: participants
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 52
participants
  No | 31
  Yes | 21

2. Primary Outcome: Best Tumor Response
Description: Response is measured according to Response Evaluation Criteria in Solid Tumors Criteria (RECIST v 1.0):
  Complete Response (CR) is disappearance of all target and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart.
  Partial Response (PR) is at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD.
  Disease Progression is at least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD or the appearance of new lesions within 8 weeks of study entry.
  Stable Disease is any condition not meeting the above criteria.
  Indeterminate is defined as having no repeat tumor assessments following initiation of study therapy for reasons unrelated to symptoms or signs of disease.
Time Frame: study entry through completion
Population: Total number eligible and evaluable participants
Measure: Number; unit: participants
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 52
participants
  Complete Response | 1
  Partial Response | 6
  Stable Disease | 26
  Disease Progression | 17
  Indeterminate | 2

3. Primary Outcome: Number of Patients With Toxicity of Bevacizumab as Assessed by CTCAE v3.0 in This Cohort of Patients.
Time Frame: Up to 5 years
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1 (CTCAE v 3.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria version 3.0
- Grade 2 (CTCAE v 3.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria version 3.0
- Grade 3 (CTCAE v 3.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria version 3.0
- Grade 4 (CTCAE v 3.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria version 3.0
- Grade 5 (CTCAE v 3.0): Number of patients who experienced a grade 5 event using Common Terminology Criteria version 3.0
Arm/Group | Grade 0 | Grade 1 (CTCAE v 3.0) | Grade 2 (CTCAE v 3.0) | Grade 3 (CTCAE v 3.0) | Grade 4 (CTCAE v 3.0) | Grade 5 (CTCAE v 3.0)
Number analyzed (Participants) | 52 | 52 | 52 | 52 | 52 | 52
Participants
  Leukopenia | 48 | 4 | 0 | 0 | 0 | 0
  Thrombocytopenia | 46 | 6 | 0 | 0 | 0 | 0
  Neutropenia | 50 | 2 | 0 | 0 | 0 | 0
  Anemia | 36 | 9 | 6 | 1 | 0 | 0
  Hypersensitivity | 50 | 1 | 1 | 0 | 0 | 0
  Rhinitis | 50 | 1 | 1 | 0 | 0 | 0
  Hypertension | 43 | 2 | 3 | 4 | 0 | 0
  Hypotension | 50 | 1 | 0 | 1 | 0 | 0
  Other Cardiac | 48 | 3 | 1 | 0 | 0 | 0
  Constitutional | 17 | 23 | 10 | 2 | 0 | 0
  Dermatologic | 47 | 5 | 0 | 0 | 0 | 0
  Nausea | 44 | 6 | 2 | 0 | 0 | 0
  Vomiting | 46 | 4 | 2 | 0 | 0 | 0
  GI | 28 | 21 | 2 | 1 | 0 | 0
  Hemorrhage | 40 | 9 | 1 | 1 | 1 | 0
  Hepatobiliary | 51 | 0 | 0 | 1 | 0 | 0
  Infection | 47 | 0 | 5 | 0 | 0 | 0
  Edema (limb) | 48 | 3 | 0 | 1 | 0 | 0
  Metabolic | 30 | 16 | 3 | 1 | 2 | 0
  Musculoskeletal | 48 | 1 | 0 | 3 | 0 | 0
  Neurosensory | 48 | 4 | 0 | 0 | 0 | 0
  Other neurologic | 47 | 4 | 0 | 1 | 0 | 0
  Ocular/visual | 49 | 3 | 0 | 0 | 0 | 0
  Pain | 33 | 11 | 4 | 4 | 0 | 0

4. Secondary Outcome: Progression-free Survival
Description: Progression is defined according to RECIST v1.0 as at least a 20% increase in the sum of LD target lesions taking as reference the smallest sum LD recorded since study entry, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or unequivocal progression of existing non-target lesions.
Time Frame: Every other cycle for the first 6 months; then every 4 cycles until progression or death, up to 5 years.
Population: Eligible and treated patients.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 52
months | 4.17 [1.38 to 8.57]

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: Every cycle during treatment, then every 3 months for the first 2 years, then every six months for the next three years and then annually for the next 5 years.
Population: Eligible and treated patients.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 52
months | 10.55 [6.60 to 24.28]

6. Secondary Outcome: Initial Performance Status
Description: Performance Status 0 = Fully active, able to carry on all pre-disease performance without restriction Performance Status 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature, e.g., light housework, office work Performance Status 2 = Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours.
Time Frame: Baseline
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 52
Participants
  Performance Status 0 | 34
  Performance Status 1 | 17
  Performance Status 2 | 1

7. Secondary Outcome: Histologic Grade
Description: G1 - Highly differentiated adenomatous carcinoma. G2 - Differentiated adenomatous carcinoma with partly solid areas. G3 - Predominantly solid or entirely undifferentiated carcinoma.
Time Frame: Baseline
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 52
Participants
  Grade 1 | 3
  Grade 2 | 12
  Grade 3 | 37

ADVERSE EVENTS:
Time Frame: from study entry up to 5 years after stopping study treatment
Arm/Group | Treatment (Bevacizumab)
Serious Adverse Events (participants affected / at risk) | 18/52
Other Adverse Events (participants affected / at risk) | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Bevacizumab) (N=52)
Lt Ventricular Systolic Dysfunction (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 1
Death No Ctcae Term - Disease Progression Nos (General disorders) | 2
Obstruction, Gi - Rectum (Gastrointestinal disorders) | 1
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Gastrointestinal - Other (Gastrointestinal disorders) | 1
Hemorrhage, Gu - Vagina (Vascular disorders) | 1
Hemorrhage/Pulmonary - Lung (Vascular disorders) | 1
Hemorrhage, Gi - Stomach (Vascular disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Proteinuria (Metabolism and nutrition disorders) | 1
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 1
Pain: Extremity-Limb (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Bevacizumab) (N=52)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 4
Rhinitis (Immune system disorders) | 4
Auditory/Ear - Other (Ear and labyrinth disorders) | 2
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 3
Neutrophils (Blood and lymphatic system disorders) | 2
Platelets (Blood and lymphatic system disorders) | 7
Leukocytes (Blood and lymphatic system disorders) | 8
Hemoglobin (Blood and lymphatic system disorders) | 24
Palpitations (Cardiac disorders) | 5
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 1
S/N Arrhythmia: Atrial Tachycardia (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 12
Lt Ventricular Systolic Dysfunction (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 2
Inr (Vascular disorders) | 1
Sweating (General disorders) | 3
Weight Gain (General disorders) | 1
Fever (General disorders) | 6
Weight Loss (General disorders) | 4
Rigors/Chills (General disorders) | 4
Fatigue (General disorders) | 38
Insomnia (General disorders) | 8
Death No Ctcae Term - Disease Progression Nos (General disorders) | 1
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 9
Bruising (Skin and subcutaneous tissue disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 8
Dry Skin (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2
Flushing (Skin and subcutaneous tissue disorders) | 1
Ulceration (Skin and subcutaneous tissue disorders) | 1
Hot Flashes (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Heartburn (Gastrointestinal disorders) | 6
Mucositis (Functional/Sympt) - Esophagus (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Distention (Gastrointestinal disorders) | 1
Taste Alteration (Gastrointestinal disorders) | 4
Dry Mouth (Gastrointestinal disorders) | 1
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 10
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 12
Anorexia (Gastrointestinal disorders) | 11
Dehydration (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 19
Diarrhea (Gastrointestinal disorders) | 17
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 2
Hemorrhage, Gu - Vagina (Vascular disorders) | 6
Hemorrhage, Gi - Rectum (Vascular disorders) | 4
Hemorrhage/Pulmonary - Respiratory Tract Nos (Vascular disorders) | 2
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 6
Hemorrhage, Gi - Anus (Vascular disorders) | 2
Hemorrhage, Gi - Oral Cavity (Vascular disorders) | 2
Hemorrhage/Bleeding - Other (Vascular disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Vein (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Otitis Media Nos (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 3
Inf Unknown Anc: Upper Airway Nos (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Vagina (Infections and infestations) | 2
Inf Unknown Anc: Mucosa (Infections and infestations) | 1
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 1
Inf Unknown Anc: Oral Cavity-Gums (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 2
Edema: Limb (Blood and lymphatic system disorders) | 7
Ast (Metabolism and nutrition disorders) | 8
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 2
Cholesterol,serum High (Metabolism and nutrition disorders) | 1
Proteinuria (Metabolism and nutrition disorders) | 5
Creatinine (Metabolism and nutrition disorders) | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 17
Ggt (Metabolism and nutrition disorders) | 1
Alt (Metabolism and nutrition disorders) | 4
Alkaline Phosphatase (Metabolism and nutrition disorders) | 9
Bilirubin (Metabolism and nutrition disorders) | 3
Lipase (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 15
Hyperuricemia (Metabolism and nutrition disorders) | 1
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 1
Amylase (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 10
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 14
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 11
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 1
Joint-Function (Musculoskeletal and connective tissue disorders) | 1
Gait/Walking (Musculoskeletal and connective tissue disorders) | 2
Cervical Spine Rom (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 4
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 2
Muscle Weakness - Extremity-Upper (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 3
Involuntary Movement (Nervous system disorders) | 1
Mood Alteration - Depression (Nervous system disorders) | 7
Mood Alteration - Anxiety (Nervous system disorders) | 7
Memory Impairment (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 5
Neuropathy-Sensory (Nervous system disorders) | 13
Neuropathy-Motor (Nervous system disorders) | 3
Ocular/Visual - Other (Eye disorders) | 3
Dry Eye (Eye disorders) | 3
Photophobia (Eye disorders) | 1
Flashing Lights/Floaters (Eye disorders) | 2
Blurred Vision (Eye disorders) | 7
Eyelid Dysfunction (Eye disorders) | 1
Pain - Other (General disorders) | 1
Pain: Pelvis (General disorders) | 3
Pain: Chest /Thorax Nos (General disorders) | 2
Pain: Chest Wall (General disorders) | 2
Pain: Head/Headache (General disorders) | 16
Pain: Neck (General disorders) | 3
Pain: Extremity-Limb (General disorders) | 9
Pain: Buttock (General disorders) | 1
Pain: Back (General disorders) | 10
Pain: Joint (General disorders) | 6
Pain: Bone (General disorders) | 2
Pain: Stomach (General disorders) | 3
Pain: Rectum (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 13
Pain: Muscle (General disorders) | 5
Pain: Neuralgia (General disorders) | 2
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 3
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17
Leak, Gu - Urethra (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Obstruction, Gu - Ureter (Renal and urinary disorders) | 1
Incontinence, Urinary (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 3
2nd Mal: Poss. Related To Cancer Rx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less